CLINICAL TRIAL: NCT05370872
Title: Efficacy of a Remotely Administered Functional Capacity Test on Return-to-work Outcomes: a Cluster Randomized Controlled Trial
Brief Title: Efficacy of a Remotely Administered Functional Capacity Test on Return-to-work Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Waterloo (Other)
Collaborators: CBI Health (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 44076
Record Dates: First submitted 2022-05-02; First posted 2022-05-12 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2022-11

CONDITIONS: Low Back Disorder; Shoulder Disease; Musculoskeletal Injury
Keywords: Functional capacity evaluation; Return to work; Functional testing; Motivational interviewing; Telehealth

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled trial. Clinicians will be randomly assigned to administer the functional testing protocol in-person (care-as-usual) or remotely (the intervention). Clients will complete the functional testing protocol based on the group assignment of the clinician to whom they were referred to.
Who Masked: Outcomes Assessor
Masking Description: The individual responsible for comparing return-to-work outcome between groups will be blind to the group assignments
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Care-as-usual (No Intervention): Clients in this group will complete functional testing in the clinic using the care-as-usual approach.
- Remote functional testing (Experimental): Clients in this group will complete functional testing using the remote functional testing approach.
  Interventions: Diagnostic Test: Remote functional testing protocol

INTERVENTIONS:
Diagnostic Test: Remote functional testing protocol — Clients in the remote functional testing protocol group will be asked to describe their functional capacity limits using a clinician guided motivational interviewing approach and will also be asked to complete a mobility screening protocol to provide the clinician with the opportunity to observe the clients natural movements.
  Arms: Remote functional testing

SUMMARY:
Currently, injured workers are required to visit a clinic, in-person, for functional testing as part of the rehabilitation and return-to-work process. The need for in-person testing has always caused problems for workers in remote areas without easy access to clinics. COVID-19 has made the problem of access to in-person clinical testing worse. Now, many injured workers can't receive functional testing due to COVID-19 related clinic closures and isolation restrictions. The investigators aim to develop and evaluate a functional testing protocol that can be delivered remotely to solve the problem of access to in-person clinic testing. A functional test that can be completed remotely, while the client remains in their home will increase access to timely testing, improve client satisfaction by removing the need for costly and time consuming travel, and will continue to help injured workers quickly recover and return to meaningful work. This research study will help to determine if return-to-work outcomes improve, or remain unchanged, when functional testing is completed remotely relative to in the clinic.

DETAILED DESCRIPTION:
Functional testing, often referred to as functional capacity evaluation (FCE) has played a longstanding role within return-to-work (RTW). The goal of an FCE is to measure an assess an individual's functional capabilities (e.g., how much can the client lift? How hard can the client push? Can the client sit for a long period of time? etc.). Historically, FCE served to measure the degree of disability (i.e., reduction in physical capability) following a workplace injury and also helped to match workers with meaningful work suited to their (adapted) functional abilities. Presently, performance-based FCE, testing requiring clients to perform movements with different weighted objects (for instance, to measure how much someone can lift), is collected at patient intake to provide a functional capacity baseline which, in turn, informs patient-centered rehabilitation programming. Not only does this FCE information help support job matching when applied at the end stages of rehabilitation (fitting clients to work based on the adapted functional capabilities), but when applied early with the rehabilitation program, FCE also provides key insights to inform patient-centred rehabilitative strategies and work hardening approaches. FCE plays a central role in supporting early and safe RTW.

However, accessing in-person, in-clinic administered functional testing to provide these important baseline insights has been a longstanding problem in remote and rural communities, a problem now amplified by clinic disruptions and temporary closures across Ontario, Canada. COVID-19 has intensified the problem of the in-person, in-clinic requirements for baseline functional testing where many injured workers are unable to access or are delayed in accessing important FCE services. The lack of patient-specific information regarding functional abilities via baseline FCE is a direct barrier to patient-centered rehabilitation and limits early and safe RTW. To address this problem, the investigators test the efficacy of a remotely administered functional testing protocol as an alternative to in-person, in-clinic baseline functional testing.

The concept of a remotely delivered baseline FCE is not new, but has been limited to subjective self-report-based methods only (e.g., asking a client how much they think they can lift). Gross et al., (2014) provide evidence that a functional interviewing-based FCE (currently deployed within the Workers' Compensation Board - Alberta, Canada system) was equivalently useful in predicting RTW outcomes relative to performance-based FCE. However, performance-based FCE elements, such as low lifting tests also remain useful for predicting RTW outcomes and provide objective insight about movement characteristics. Observing how a client moves when performing a lift, for example, provides insight into their willingness to engage, any guarding behaviours they may exhibit, any observed hesitancy to move, and also provides insight into their coordination of movement. These insights are necessary to inform patient centered rehabilitation programming and to ensure that the care team has the necessary health professionals (i.e., rehabilitation to address mechanical issues relative to psychosocial barriers). The investigators believe that a hybrid FCE including self-report to estimate maximum functional levels combined with a safe, submaximal performance-based FCE to assess movement characteristics can provide key insights to best optimize early and safe RTW when using virtual FCE delivery. However, at present, no such testing paradigm exists.

To optimize remote FCE service delivery to include both self-report and performance-based insights, the investigators aim to leverage the 2D video recording capabilities of Microsoft Teams, the CBI Health approved software application for safely and securely engaging with clients remotely. The investigators have demonstrated how movement data (which can be generated using 2D video and pose estimation) and advances in computer vision can be leveraged to generate insightful information about key movement characteristics, functional capabilities and safety. The ability for a patient to record their performance of safe, standardized, sub-maximal actions will generate essential and objective information to support patient-centered rehabilitative programing, an integral requirement for early and safe RTW.

The investigators have developed an evidence-based protocol for remote delivery of baseline functional testing for injured workers inclusive of performance-based and self-report FCE measures. The investigators now aim to evaluate if a remotely administered functional testing protocol can generate treatment recommendations and RTW outcomes that are consistent with the current status quo requiring in-person, in-clinic functional assessment. The investigators hypothesize that the remotely administered functional testing protocol will yield similar insight to in-person, in-clinic baseline FCE, such that RTW outcomes will be equal to or better when using the remotely administered functional testing protocol. The investigators also hypothesize that patient experience and satisfaction will be improved with the use of a remotely administered functional testing protocol because time and cost intensive travel barriers can be removed.

ELIGIBILITY:
Inclusion Criteria:

* Injured workers with accepted Workplace Safety and Insurance Board (WSIB) of Ontario claims referred to CBI Health for WSIB Specialty Programs related to musculoskeletal injuries of either Back and Neck, or Upper Extremity.

Exclusion Criteria:

* Under the age of 18 years,
* referred for surgery during the time of the rehabilitation programming,
* have a concurrent traumatic brain injury or mental health disorder that takes precedence over the musculoskeletal injury, or
* require the assistance of an interpreter to read, write or speak English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Return to work recommendation at intake | Baseline measure - a intake into the rehabilitation program
  When referred to an musculoskeletal program of care, clients are classified into return to work categories based on their ability to meet job requirements as measured by the clinician using the functional testing protocol. The return to work recommendation at intake is used to inform the rehabilitation program.
Return to work recommendation at discharge | At program discharge (approximately 8-12 weeks post intake, where each client will receive a tailored program based on their return to work recommendation at intake)
  Once the client has completed a musculoskeletal program of care, clients are again classified into return to work categories based on their ability to meet job requirements as measured by the clinician using the functional testing protocol. The return to work recommendation at discharge is used to inform how the client is reintegrated into their workplace.
Return to work status | three-months post discharge
  Clients will be aske to describe their current work status at three-months post discharge by selecting 1 of 5 options (work regular, full time duties; work regular, part time duties, work light duty or modified position full time; work light duty or modified position part time; not currently working)

SECONDARY OUTCOMES:
Adverse events | Through study completion, and average of 1 year
  Reports of adverse events for participating clients will be extracted from the occupational health & safety document management system.
Client experience and satisfaction | one-week post initial functional testing session
  Clients will complete a web survey inclusive of 3 questions that probe their experience and satisfaction with the functional testing that they received. Each question is posed using a 5-point Likert scale (strongly disagree, disagree, neither agree or disagree, agree, strongly agree).

CONTACTS AND LOCATIONS:
Overall Officials: Steve Fischer, Principal Investigator — Associate Professor, University of Waterloo
Locations (5):
- Canada (5):
  - CBIH London Dundas, London, Ontario
  - CBIH London Fanshawe, London, Ontario
  - CBIH London Wonderland, London, Ontario
  - CBIH Nepean, Nepean, Ontario
  - CBIH St. Laurent, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers.

REFERENCES:
- [Result] Gross DP, Asante AK, Miciak M, Battie MC, Carroll LJ, Sun A, Mikalsky M, Huellstrung R, Niemelainen R. A cluster randomized clinical trial comparing functional capacity evaluation and functional interviewing as components of occupational rehabilitation programs. J Occup Rehabil. 2014 Dec;24(4):617-30. doi: 10.1007/s10926-013-9491-4. PMID 24374369